CLINICAL TRIAL: NCT00553813
Title: A Phase 2, Open Label, Single Arm Trial of TPI 287 in Patients With Advanced, Unresectable Pancreatic Cancer After Prior Treatment With a Gemcitabine-based Therapy
Brief Title: A Phase II Trial of TPI 287 in Patients Advanced, Unresectable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPI 287-06
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Pancreatic Cancer
Keywords: Unresectable; Gemcitabine; Taxane; TPI 287
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — TPI-287

INTERVENTIONS:
Drug: TPI 287 — Intravenous dose of 125 mg/m2 TPI 287 on Day 1, Day 8, and Day 15 in a repeating 28 day cycle.

SUMMARY:
The primary objective of the study is to assess the activity of TPI 287 as single agent therapy for patients with advanced, unresectable pancreatic cancer after failure of gemcitabine-containing therapy. Activity of TPI 287 will be determined by the 6-month survival rate.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single arm Phase 2 study in patients with advanced, unresectable pancreatic cancer who have received prior gemcitabine-based chemotherapy for their disease. Patients will receive TPI 287 administered as a 60-minute (± 10 min) IV infusion.

The primary endpoint of the trial will be the 6-month survival rate. Additional efficacy endpoints will be response rate, duration of response and stable disease, and 6-month progression free survival. Responses will be assessed by reduction in radiographically measurable disease as defined by the RECIST criteria. Time to worsening of clinical status will be based on reductions in pain and/or analgesic use and changes in tumor markers (CA 19-9) will also be followed.

Patients will remain on study until tumor progression or death, unacceptable toxicity, withdrawal of consent or discontinuation based on Investigator discretion. Patients will be followed for survival for up to 1 year after enrollment on the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological confirmation of ductal adenocarcinoma or undifferentiated carcinoma of the pancreas
* Patients must have metastatic disease precluding curative surgery
* Patients must have received only one prior systemic anticancer treatment for their advanced disease, which must have included a gemcitabine-based therapeutic regimen for advanced disease
* Patients may have received prior adjuvant therapy for their disease
* Patients must have a Karnofsky performance status ≥ 70 (Appendix I)
* Patients must be ≥ 18 years of age
* Women of childbearing potential (WOCBP):

  * Must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study
  * Must have a negative serum or urine pregnancy test
* Patients must have adequate organ function:

  * Bone marrow reserve as evidenced by: Absolute neutrophil count ≥1,500/uL, Platelet count ≥ 100,000/uL
  * Renal function as evidenced by serum creatinine ≥ 2.0 mg/uL
  * Hepatic function as evidenced by: Serum total bilirubin < 2.0 mg/uL, SGOT/SGPT < 3X ULN for the reference lab (< 5X ULN for patients with known hepatic metastases)
* Patient must have recovered from prior surgery, radiotherapy or other antineoplastic therapy
* Patients or their legal representative must be able to read, understand, and sign the informed consent to participate in the trial

Exclusion Criteria:

* Patients with islet cell tumors, lymphoma, or sarcoma of the pancreas
* Patients with more than one prior treatment for metastatic pancreatic carcinoma
* Patients with current peripheral neuropathy > Grade 1
* Patients receiving any concurrent chemotherapy, radiotherapy, hormonal therapy or immunotherapy
* Patients with serious infection or a life-threatening illness (unrelated to tumor) that is > Grade 2 NCI CTCAE V 3.0), or active, serious infections requiring parental antibiotic therapy within 4 weeks prior to screening
* History of cardiac disease or events according to the New York Health Association (NYHA) assessments. Clinically evident congestive heart failure as defined by NYHA Class 3 or 4 CHF or cardiac arrhythmia, including atrial fibrillation, if not adequately controlled
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results
* Known HIV or Hepatitis B or C (active, previously treated or both)
* A history of other malignancy (except nonmelanoma skin cancer or carcinoma-in-situ of cervix), unless in CR and not receiving therapy for that disease for a minimum of 5 years
* Patients with known hypersensitivity to any of the components of the drugs to be administered on study
* Patients receiving concurrent investigational therapy (investigational therapy is defined as treatment for which there is currently no regulatory authority-approved indication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Survival | 6 Months

SECONDARY OUTCOMES:
Overall Response Rate | Ongoing
Evaluate time to worsening of clinical status as measured by changes in pain, Karnofsky score, and weight. | Ongoing
Response rates and time to progression of tumor marker levels (CA 19-9) | Ongoing
Assess the safety and tolerability of TPI 287 in this patient population | Ongoing
Evaluate outcomes of patient subsets defined by duration of prior gemcitabine therapy | Ongoing
Evaluate the gene expression profile in relation to clinical outcomes | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Silberman, MD, Study Director — SLS Oncology, LLC
Locations (4):
- United States (3):
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Sidney Kimmel Comprehensive Cancer Center - Johns Hopkins University, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
- Hospital Madrid, Madrid, Spain